CLINICAL TRIAL: NCT00057174
Title: Economic Impact of Guidelines for Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 99-238
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Gastroesophageal Reflux Disease; Health Economics
Keywords: Proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Disease management of gastroesophageal reflux disease

INTERVENTIONS:
Drug: Disease management of gastroesophageal reflux disease

SUMMARY:
This is a series of two prospective studies based on the Department of Veterans Affairs drug treatment guideline for the pharmacologic management of gastroesophageal reflux disease. Our hypothesis is that novel strategies for medical management of gastroesophageal reflux disease (GERD) can decrease resource utilization without adversely affecting patient quality of life. The strategies tested in this project included 1) step-down management, whereby patients rendered asymptomatic on proton pump inhibitors (PPIs) are treated with less expensive medication, and 2) intermittent therapy, defined as administration of medication only for recurrence of GERD symptoms. We chose to examine an intermittent strategy of PPI administration since in addition to the VA guideline requiring step-down therapy, over-the-counter PPIs administered by intermittent therapy became available for use by patients during the study period.

DETAILED DESCRIPTION:
Background:

This is a series of two prospective studies based on the Department of Veterans Affairs drug treatment guideline for the pharmacologic management of gastroesophageal reflux disease. Our hypothesis is that novel strategies for medical management of gastroesophageal reflux disease (GERD) can decrease resource utilization without adversely affecting patient quality of life. The strategies tested in this project included 1) step-down management, whereby patients rendered asymptomatic on proton pump inhibitors (PPIs) are treated with less expensive medication, and 2) intermittent therapy, defined as administration of medication only for recurrence of GERD symptoms. We chose to examine an intermittent strategy of PPI administration since in addition to the VA guideline requiring step-down therapy, over-the-counter PPIs administered by intermittent therapy became available for use by patients during the study period.

Objectives:

The objectives of this project are to determine the efficacy of step-down therapy and intermittent therapy in patients with GERD, and the impact of these strategies on direct healthcare costs and health-related quality of life (HRQOL). Additionally, we will examine patient factors predictive of non-response to these management strategies that may be alternatives to traditional continuous PPI administration.

Methods:

Two separate studies were conducted in our population of patients with GERD symptoms (heartburn or acid regurgitation) rendered asymptomatic on PPIs. Both studies randomized subjects to an intervention strategy (Step-down or Intermittent therapy) or to a control group in which PPIs were continued on a daily basis.

Step-down therapy: Step-down subjects discontinued PPIs and were prescribed histamine2-receptor antagonists (H2RAs) for 2 weeks, and if still asymptomatic, H2RAs were discontinued. If symptoms recurred, H2RAs were reinitiated, and if still symptomatic, subjects were prescribed PPIs at the dose that initially alleviated their symptoms. Intermittent therapy: Intermittent therapy subjects discontinued daily use of PPIs and were prescribed short courses of PPI (daily for 8 weeks) for recurrence of GERD symptoms. The primary efficacy measure was the proportion of subjects remaining free of GERD symptoms while on their prescribed therapy (step-down group: no symptoms on H2RAs or no GERD medication; intermittent therapy group: no PPIs for �2 weeks after discontinuation, and < 3 symptom recurrences requiring PPIs; control groups: no GERD symptoms on PPI). Follow up was conducted for 6 months after randomization. In addition to the primary efficacy measure, we examined total resource utilization (pharmacy and non-pharmacy), HRQOL, and potential predictors of non-response to step-down or intermittent therapy (requirement of daily PPI to control symptoms). Logistic regression and random-effects models adjusted for covariates and clustering effects.

Status:

Enrollment and follow-up have been completed. Efficacy measures are reported above. Outcome measures including comparison of direct health care costs, health-related quality of life, and determinants of non-response to step-down or intermittent therapy are being examined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with GERD symptoms treated with PPIs. For the purpose of this study, GERD symptoms include heartburn or acid regurgitation. Symptoms of dyspepsia (epigastric pain, nausea, bloating, early satiety) may be present, but may not be used as the sole criteria for inclusion into the study.
2. Asymptomatic (no heartburn or acid regurgitation) on PPI therapy.

Exclusion Criteria:

1. Complications of gastroesophageal reflux disease including esophageal stricture, hemorrhage due to erosive esophagitis, Barrett�s esophagus or adenocarcinoma of the esophagus, or extra-esophageal manifestations of reflux disease (pulmonary or laryngeal disease due to acid reflux).
2. Concurrent diagnoses of other gastrointestinal diseases including gastric or duodenal ulcer, Zollinger-Ellison syndrome or other hypersecretory disorders, or gastric cancer.
3. Esophagitis secondary to non-acid peptic causes: infections (viral, bacterial, fungal), or medications causing esophageal erosions.
4. Inability to maintain follow-up, either due to excessive distance to the VA primary care facility or lack of telephone services.
5. Unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Inadomi, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] El-Serag HB, Graham DY, Richardson P, Inadomi JM. Prevention of complicated ulcer disease among chronic users of nonsteroidal anti-inflammatory drugs: the use of a nomogram in cost-effectiveness analysis. Arch Intern Med. 2002 Oct 14;162(18):2105-10. doi: 10.1001/archinte.162.18.2105. PMID 12374519
- [Result] Rubenstein JH, Inadomi JM. Empiric beta-blockers for the prophylaxis of variceal hemorrhage: cost effective or clinically applicable? Hepatology. 2003 Feb;37(2):249-52. doi: 10.1053/jhep.2003.50089. No abstract available. PMID 12540773
- [Result] Rubenstein JH, Inadomi JM. Dysphagia drives doctors to diagnose a disease: pitfalls in interpreting observational studies. Gastrointest Endosc. 2005 Jun;61(7):809-11. doi: 10.1016/s0016-5107(05)00544-4. No abstract available. PMID 15933680
- [Result] Rubenstein JH, Vakil N, Inadomi JM. The cost-effectiveness of biomarkers for predicting the development of oesophageal adenocarcinoma. Aliment Pharmacol Ther. 2005 Jul 15;22(2):135-46. doi: 10.1111/j.1365-2036.2005.02536.x. PMID 16011672
- [Result] Rubenstein JH, Davis J, Marrero JA, Inadomi JM. Relationship between diabetes mellitus and adenocarcinoma of the oesophagus and gastric cardia. Aliment Pharmacol Ther. 2005 Aug 1;22(3):267-71. doi: 10.1111/j.1365-2036.2005.02544.x. PMID 16091065
- [Result] Rhee J, Scheiman J, Inadomi J. "Spontaneous" passage of a pancreatic duct stone. Gastrointest Endosc. 2003 Feb;57(2):278-80. doi: 10.1067/mge.2003.62. No abstract available. PMID 12556808
- [Result] Chey WD, Inadomi JM, Booher AM, Sharma VK, Fendrick AM, Howden CW. Primary-care physicians' perceptions and practices on the management of GERD: results of a national survey. Am J Gastroenterol. 2005 Jun;100(6):1237-42. doi: 10.1111/j.1572-0241.2005.41364.x. PMID 15929751
- [Result] Inadomi JM, Jamal R, Murata GH, Hoffman RM, Lavezo LA, Vigil JM, Swanson KM, Sonnenberg A. Step-down management of gastroesophageal reflux disease. Gastroenterology. 2001 Nov;121(5):1095-100. doi: 10.1053/gast.2001.28649. PMID 11677201
- [Result] Inadomi JM, McIntyre L, Bernard L, Fendrick AM. Step-down from multiple- to single-dose proton pump inhibitors (PPIs): a prospective study of patients with heartburn or acid regurgitation completely relieved with PPIs. Am J Gastroenterol. 2003 Sep;98(9):1940-4. doi: 10.1111/j.1572-0241.2003.07665.x. PMID 14499769
- [Result] Inadomi JM. Update on the cost-effectiveness of screening for colorectal neoplasia. Curr Opin Gastroenterol. 2003 Jan;19(1):44-50. doi: 10.1097/00001574-200301000-00008. PMID 15699893
- [Result] Inadomi JM. On-demand and intermittent therapy for gastro-oesophageal reflux disease: economic considerations. Pharmacoeconomics. 2002;20(9):565-76. doi: 10.2165/00019053-200220090-00001. PMID 12141885
- [Result] Inadomi JM, Sampliner R, Lagergren J, Lieberman D, Fendrick AM, Vakil N. Screening and surveillance for Barrett esophagus in high-risk groups: a cost-utility analysis. Ann Intern Med. 2003 Feb 4;138(3):176-86. doi: 10.7326/0003-4819-138-3-200302040-00009. PMID 12558356
- [Result] Inadomi JM. Cost-effectiveness of colorectal cancer surveillance in ulcerative colitis. Scand J Gastroenterol Suppl. 2003;(237):17-21. doi: 10.1080/00855910310001430. PMID 12797675
- [Result] Inadomi JM, Fendrick AM. PPI use in the OTC era: who to treat, with what, and for how long? Clin Gastroenterol Hepatol. 2005 Mar;3(3):208-15. doi: 10.1016/s1542-3565(04)00717-7. PMID 15765438
- [Result] Inadomi J, Fendrick AM. Dyspepsia: Physicians Information and Education Resource. PIER. 2003 Jan 1.
- [Result] Cram P, Fendrick AM, Inadomi J, Cowen ME, Carpenter D, Vijan S. The impact of a celebrity promotional campaign on the use of colon cancer screening: the Katie Couric effect. Arch Intern Med. 2003 Jul 14;163(13):1601-5. doi: 10.1001/archinte.163.13.1601. PMID 12860585